CLINICAL TRIAL: NCT06873126
Title: A Two-group Experimental Trial to Promote Sports and Exercise Among Female University Students in Saudi Arabia: the Relationship Between Mental Health and Adherence to Phyicsal Activity
Brief Title: Two Group Experimental Trial Promoting Sports and Exercise Among Female University Students in Saudi Arabia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Vandana Esht, Associate Professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC-46/06/1229
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mental health (Active Comparator): To compare the relationship between mental health and adherence to physical activity
  Interventions: Combination Product: Counselling sessions
- Physical activity (Active Comparator): To compare the relationship between mental health and adherence to physical activity
  Interventions: Combination Product: Counselling sessions

INTERVENTIONS:
Combination Product: Counselling sessions — The study provides insights into the use of awareness counselling sessions for physical activity promotion, which may have a significant impact on physical activity education, promotion, practice and policy making and will be more effective to ensure adherence to activity among young adults.

SUMMARY:
The study provides insights into the use of awareness counselling sessions for physical activity promotion, which may have a significant impact on physical activity education, promotion, practice and policy making and will be more effective to ensure adherence to activity among young adults.

ELIGIBILITY:
Inclusion Criteria:

* Participants scoring between 0 to 10 (normal) and 11 to 16 (mild) and 16 to 20 (moderate) in DASS-21 depression subscale
* voluntary participants
* physical activity level lightly active

Exclusion Criteria:

* University students diagnosed with psychiatric disorders and taking therapy or family history of mental illness
* Students with comorbid conditions such as chronic pain, respiratory disorders, musculoskeletal diseases, cardiac diseases, neurological diseases or any disabilities and pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
daily moderate- to vigorous-intensity physical activity (MVPA), physical activity level (PAL) evaluated using IPAQ-SF | 7 days
  International Physical Activity Questionnaire Short Form (IPAQ-SF) was used to measure the physical activity among students. The IPAQ measures the type and intensity of physical activity and time spent walking and sitting in a duration of 7 days. A higher IPAQ score indicates a higher intensity of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Jizan, Jazan Region, Saudi Arabia